CLINICAL TRIAL: NCT07041567
Title: THE EFFECT OF LOW-FLOW-ANESTHESİA ON POSTOPERATİVE ATELECTASİS İN PATİENTS UNDERGOİNG BARİATRİC SURGERY: AN EVALUATİON USİNG ULTRASOUND
Brief Title: İn This Study, Patients Undergoing Bariatric Surgery Will be Divided Into Two Groups. The Control Group Will Receive Normal-flow, While the Study Group Will Receive Low-flow Inhalational Anesthesia. The Aim is to Compare the Incidence of Postop Atelectasis-between the Two Groups Using USG Evaluation
Acronym: BCAİA-AUD28
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Dunyakhanim Farzaliyeva, RESIDENT DOCTOR, Goztepe Prof Dr Suleyman Yalcın City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: BCAİA-AUD28
Record Dates: First submitted 2025-06-16; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Atelectasis; Pulmonary Complications; Ultrasonography
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (group N) - Standard flow anesthesia (Active Comparator): İnhalational anesthesia
  Interventions: Other: Inhalational anesthesia
- İntervention group (Group D) - Low Flow Anesthesia (Experimental): İnhalational anesthesia
  Interventions: Other: Inhalational anesthesia

INTERVENTIONS:
Other: Inhalational anesthesia — In Group D, patients undergoing bariatric surgery will receive low-flow inhalational anesthesia (0.5-1 L/min) with sevoflurane. The aim is to evaluate whether the reduced fresh gas flow rate decreases the incidence of postoperative atelectasis, assessed via pulmonary ultrasonography.
  In Group N, patients undergoing bariatric surgery will receive standard-flow inhalational anesthesia (2-4 L/min) with sevoflurane. This group serves as the comparator to evaluate the impact of flow rate on postoperative atelectasis incidence.
  Other Names: Normal flow inhalational anesthesia (Group N); Low flow inhalational anesthesia (Group D)

SUMMARY:
This study is a clinical trial and its purpose is to evaluate the effect of low and normal flow anesthesia on atelectasis formation in patients undergoing bariatric surgery by ultrasonography.

In this study, lung ultrasounds and respiratory function tests will be performed on volunteers before and after surgery. These procedures are completely painless and safe.

No invasive procedure will be performed in the study; the methods used do not pose any additional risk other than existing treatment procedures.

ELIGIBILITY:
Inclusion Criteria:

* Will undergo Sleeve Gastrectomy surgery;
* 18-65 years old
* ASA III patients.

Exclusion Criteria:

* Patients who do not give consent
* Patients with ASA 4 and above
* Those with serious respiratory comorbidities (interstitial lung disease, serious permanent lung diseases)
* Uncontrolled Hypertension, Diabetes Mellitus
* Under 18 and over 65 years of age
* Chronic renal failure, Liver failure
* CHF (EF<30) will not be included in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-20 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
the atelectasis rate with the Lung Ultrasound score (AUS score). | 8 months